CLINICAL TRIAL: NCT00920556
Title: A Phase II, Open-Label, Clinical Study to Assess the Safety and Activity of SRT501 Alone or in Combination With Bortezomib in Patients With Multiple Myeloma
Brief Title: A Clinical Study to Assess the Safety and Activity of SRT501 Alone or in Combination With Bortezomib in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated.24 subjects enrolled;provided adequate data for decision making.
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113222
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Resveratrol; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): 5.0 g SRT501 will be administered for 20 consecutive days in a 21 day cycle for a maximum of 12 cycles. SRT501 will be administered at the same time each morning (approximately 15-30 minutes after breakfast) on all dosing days. No SRT501 administration will occur on Day 21 of each cycle.
  After the first two cycles of SRT501, any subject who exhibits stable disease or better with SRT501 monotherapy (5.0 g/day) will continue for an additional two cycles. If, after the first two cycles, a subject exhibits PD, that subject will receive bortezomib (1.3 mg/m2 on Day 1, Day 4, Day 8, and Day 11 in a 21 day cycle) in conjunction with SRT501. Bortezomib will be administered prior to breakfast and SRT501 administration.
  If after two additional cycles of SRT501 monotherapy (4 cycles total), the subject exhibits a MR or better, they they will remain on SRT501 therapy. If PD or SD are exibited, they are to undergo bortezomib regiment listed above.
  Interventions: Drug: 5.0g SRT501; Drug: Bortezomib

INTERVENTIONS:
Drug: 5.0g SRT501 — 5.0g SRT501 will be supplied in clinical kits as a powder which will be reconstituted with vehicle and water into a liquid suspension. SRT501 will be administered orally as a liquid suspension for 20 consecutive days in each 21 day cycle.
Drug: Bortezomib — Bortezomib (1.3 mg/m2) will be given as an intravenous solution in a 3-5 second push on Day 1, 4, 8 and 11 in every 21 day cycle.

SUMMARY:
The primary purpose of this study is to determine the safety and tolerability of SRT501 (5.0 g) with or without concurrent bortezomib administration, when administered once daily in 21 day cycles, in male and female subjects with Multiple Myeloma.

The purpose is also to define objective response (ORR, CR, PR, MR, SD) and time to progression (TTP) of SRT501 with or without concurrent bortezomib administered concurrently in male and female subjects with Multiple Myeloma.

In addition, 15 subjects will participate in a sub-study to assess the pharmacokinetics of SRT501.

DETAILED DESCRIPTION:
This is an, open-label, phase II study of SRT501, alone or in combination with bortezomib, in subjects with measurable Multiple Myeloma. Sixty-one (61) evaluable subjects, who fulfill the inclusion/exclusion criteria, will be enrolled in this study. Pharmacokinetic (PK) samples will be collected from a subset of 15 subjects to determine SRT501 plasma concentrations in this patient population. Subjects will sign the informed consent form prior to any study related procedures. If eligible, subjects will receive 5.0 g of SRT501 to be administered for 20 consecutive days in a 21 day cycle for a maximum of 12 cycles. SRT501 will be administered as an oral suspension product at the same time each morning (approximately 15-30 minutes following consumption of breakfast) on all dosing days. Safety assessments will be performed continuously throughout the cycle and these will be reviewed for all subjects at Day 21 of each cycle prior to subjects proceeding to the next cycle. SRT501 will not be administered on Day 21 of each cycle. Subjects will be assessed for efficacy and response of SRT501 at the end of every 2 cycles (6 weeks) of treatment. When necessary, a bone marrow biopsy and CT (or appropriate radiographic imaging) of the chest and abdomen/pelvis will be performed to confirm response. After the first two cycles of SRT501 treatment and review of the efficacy and response analysis, any subject who exhibits stable disease or better with SRT501 monotherapy may continue on SRT501 monotherapy (5.0 g/day) for an additional two cycles. If, after the first two cycles of SRT501 monotherapy, a subject exhibits PD, then that subject will receive bortezomib (1.3 mg/ m2 on Day 1, Day 4, Day 8, and Day 11 in a 21 day cycle) in conjunction with SRT501 (5.0 g/day). Bortezomib will be administered prior to SRT501 administration. If after two additional cycles of SRT501 monotherapy (4 cycles total), the subject exhibits a MR or better, they will remain on SRT501 (5.0 g/day) treatment until they are judged to have SD or PD. At the time the subject is judged to have SD or PD after receiving at least four cycles of SRT501 (5.0 g/day) monotherapy, then they may also receive bortezomib (1.3 mg/m2 on Day 1, Day 4, Day 8, and Day 11 in a 21 day cycle) in conjunction with daily SRT501 dosing. If at any point while a subject is receiving SRT501 and bortezomib the subject is assessed to have PD, then they will be removed from the study and will be required to undergo End of Study assessments/follow-up approximately 28 days (+/- 7 days) following the last dose of SRT501 or SRT501 and bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be male or female ≥ 18 years at the time of signing Informed Consent.
* Subject was previously diagnosed with Multiple Myeloma and has failed at least one prior treatment regimen for the disease.
* Subject must have measurable disease.
* Subjects must have relapsed or relapsed/refractory disease as defined in Appendix 4.
* Subject must have a life expectancy of greater than 6 months.
* Subject has an ECOG Performance status of 0 to 2 (Appendix 2).
* Subject has no prior history of HIV-1, HIV-2, Hepatitis B or C infection.
* Subject has a normal 12 lead ECG or an ECG with an abnormality considered to be clinically insignificant.
* Subject has the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described.
* Subject must be able to adhere to the study visit schedule and other protocol requirements.
* Subject must understand and voluntarily sign an informed consent document.
* All subjects of reproductive potential must agree prior to study entry to use adequate contraception (hormonal or double barrier method of birth control; abstinence) for the duration of the study dosing and at least 12 weeks after completion of study drug.
* Adequate end organ function, defined as the following:

  * Total bilirubin < 2 x ULN, unless attributable to Gilbert's disease
  * ALT (SGPT) and AST (SGOT) < 2.5 x ULN
  * Creatinine < 2.0 x ULN
  * ANC > 0.5 x 10^9/L
  * Platelets > 20,000 cells/mm3

Exclusion Criteria:

* Intolerance to resveratrol, SRT501 or bortezomib or significant allergy to either compound, boron or mannitol or significant prior toxicity with either agent that would preclude the safe use of that agent. Prior therapy with either compound is permitted.
* Subjects with other active malignancy, with the exception of basal cell or squamous cell carcinoma of the skin.
* An uncontrolled intercurrent illness including, but not limited to, recent (≤ 6 months), ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, acute diffuse infiltrative pulmonary or pericardial disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject with a history of or current gastro-intestinal diseases influencing drug absorption, with the exception of an appendectomy.
* Women who are breast-feeding, pregnant, expect to become pregnant during the course of the study, or are sexually active in a heterosexual relationship and are not using a medically acceptable double barrier method birth control. Confirmation that the subject is not pregnant must be established by a negative serum beta-hCG pregnancy test result obtained during the Screening period. Pregnancy testing is not required for post-menopausal or surgically sterilized women. Women relying solely on oral contraceptives for birth control are excluded.
* Subjects who have had chemotherapy or radiotherapy within 4 weeks prior to signing Informed Consent or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Subjects who are on any concurrent medications that may exhibit anti-neoplastic therapy, with the exception of < 10 mg of prednisone or equivalent as indicated for other medical conditions, or up to 100 mg of hydrocortisone as premedication for administration of certain medications or blood products.
* Subjects currently taking any investigational therapies and/or dietary supplements containing resveratrol.
* Subjects with peripheral neuropathy of Grade 2 or greater.
* Subjects with uncontrolled bleeding.
* Subjects with evidence of mucosal or internal bleeding and/or platelet refractory (i.e., unable to maintain a platelet count ≥ 20,000 cells/mm3).
* Subjects with a hemoglobin < 8.0 g/dL. Transfusions and/or EPO treatment are permitted in subjects who are potentially excluded by this criteria.
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator, would preclude treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03-30 (Actual); Primary Completion 2010-11-04 (Actual); Study Completion 2010-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Vejle, Denmark
- United Kingdom (4):
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Popat R, Plesner T, Davies F, Cook G, Cook M, Elliott P, Jacobson E, Gumbleton T, Oakervee H, Cavenagh J. A phase 2 study of SRT501 (resveratrol) with bortezomib for patients with relapsed and or refractory multiple myeloma. Br J Haematol. 2013 Mar;160(5):714-7. doi: 10.1111/bjh.12154. Epub 2012 Dec 4. No abstract available. PMID 23205612
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113222 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113222 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113222 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113222 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113222 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113222 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants with Multiple Myeloma were enrolled in the study. The study was conducted at four centers in United Kingdom and 1 center in Denmark, and was terminated early.
Groups:
- Overall Study: Eligible participants were administered 5 gram (g) of SRT501, as oral suspension every morning approximately 15-30 minutes after breakfast), for 20 days in 21-day cycle, for max period of 12 cycles (Not administered on Day 21 of each cycle). Post first two cycles, participant who exhibited stable disease (SD) or better, with SRT501 monotherapy, continued for additional two cycles. If, after first 2 cycles, participant exhibited PD, then received bortezomib (1.3 milligram(mg)/meter square (m^2)on Day 1, Day 4, Day 8, and Day 11 in a 21 day cycle) along with SRT501. Bortezomib was administered intravenous suspension, prior to breakfast and SRT501 administration. If after 2 additional cycles of SRT501 monotherapy (4 cycles total), participant exhibited SD or better, they remained on SRT501 therapy, until judged to have PD. If PD,participants underwent bortezomib regiment as above. At any point of (SRT501+Bortezoimb),participant was assessed with PD, was discontinued
Period: Overall Study
Arm/Group | Overall Study
Started | 24
Completed | 0
Not Completed | 24
Not completed — Adverse Event | 16
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Eligible participants were administered 5 gram (g) of SRT501, as oral suspension every morning approximately 15-30 minutes after breakfast), for 20 days in 21-day cycle, for max period of 12 cycles (Not administered on Day 21 of each cycle). Post first two cycles, participant who exhibited stable disease (SD) or better, with SRT501 monotherapy, continued for additional two cycles. If, after first 2 cycles, participant exhibited progressive disease (PD), then received bortezomib (1.3 milligram(mg)/meter square (m^2)on Day 1, Day 4, Day 8, and Day 11 in a 21 day cycle) along with SRT501. Bortezomib was administered intravenous suspension, prior to breakfast and SRT501 administration. If after 2 additional cycles of SRT501 monotherapy (4 cycles total), participant exhibited SD or better, they remained on SRT501 therapy, until judged to have PD. If PD,participants underwent bortezomib regiment as above. At any point of (SRT501+Bortezoimb),participant was assessed with PD, was discontinued
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Afro-Caribbean | 3
  Race: Caucasian | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, or is an important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or a drug-induced liver injury.
Time Frame: Approximately up to 12 cycles of 3 weeks each
Population: Safety Population was defined as all the participants who received any amount of SRT501 or bortezomib.
Measure: Count of Participants; unit: Participants
Groups:
- SRT501 Monotherapy: The eligible participants in this arm received 5 g of SRT501, oral suspension every morning at the same time approximately 15-30 minutes following consumption of breakfast) on all dosing days, for 20 consecutive days in a 21-day cycle for a maximum period of 12 cycles. There was no time between the cycles i.e Day 1 of a cycle was started on the day following Day 21 of the previous cycle. SRT501 was not administered on Day 21 of each cycle.
- SRT501 + Bortezomib: The eligible participants in this arm received an intravenous solution of Bortezomib at 1.3 mg/m^2 in conjunction with SRT501 (5.0 g/day) daily dosing. Bortezomib was administered prior to breakfast and SRT501 administration, on Day 1, 4, 8 and 11 in every 21 day cycle. It was given as per the local institution's guidelines and standards of care. SRT501 + Bortezomib, is a subset of arm SRT501 monotherapy.
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 24 | 9
Participants
  Any AE | 24 | 9
  Any SAE | 12 | 3

2. Primary Outcome: Number of Participants With Overall Response Rate
Description: Overall response rate, defines proportion of participants with Complete response (CR), Partial response (PR) or Minimal response (MR) as best response for all cycles. In atleast 2 determinations for minimum of 6 week (Wks) for every criteria listed. CR defined as disappearance of original monoclonal (MC) paraprotein (PP) in blood and urine on immunofixation determinations (IFD); < 5 % plasma cells in bone marrow; no increase in size or number of lytic bone lesions (LBLs); disappearance of soft tissue plasmacytomas (STP). PR defined as >= 50% reduction (RE) in level of serum MC PP for 2 IFDs; if present RE in 24 hour urinary light chain excretion (ULCE) by >= 90% RE or <200 mg; >= 50% RE in STP for; no increase in size or number of LBLs. MR criteria defined were >= 25% to <=49% RE serum MC PP; if present 50 to 89% RE in 24 hour LCE exceeding 200 mg/24 hour; 25% to 49% RE in size of STP; no increase in size or number of LBLs.
Time Frame: Approximately up to 12 cycles of 3 weeks
Population: Modified Intent to Treat (mITT), had participants who completed first (2) cycles of SRT501 monotherapy. Participants dropped were not counted; those withdrew after 2nd cycle were considered evaluable regardless of discontinuation reason; alongwith participants discontinued for missing clinical trial material after 2 cycle, were considered.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 0 | 3

3. Primary Outcome: Number of Participants With Partial Response (PR) as Best Response (BR)
Description: PR includes some, but not all, criteria for CR providing the remaining criteria are satisfied: ≥50% reduction in the level of serum monoclonal paraprotein for at least 2 immunofixation determinations for a minimum of 6 weeks, If present, reduction in 24 hr urinary light chain excretion by either ≥90% or to <200 mg for at least 2 determinations for a minimum of 6 weeks, ≥50% reduction in the size of soft tissue plasmacytomas (by clinical or radiographic examination) for a minimum of 6 weeks, No increase in size or number of lytic bone lesions (development of compression fracture does not exclude response).
Time Frame: Up to 12 cycles of 3 weeks each
Population: mITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 0 | 2

4. Primary Outcome: Number of Participants With Minor Response (MR) as Best Response (BR)
Description: MR includes some, but not all, criteria for PR providing the remaining criteria satisfied: ≥25% to ≤ 49% reduction in the level of serum monoclonal paraprotein for at least 2 immunofixation determinations for a minimum of 6 weeks, If present, a 50 to 89% reduction in 24 hr light chain excretion, which still exceeds 200 mg/24 hr, for at least 2 determinations for a minimum of 6 weeks, 25-49% reduction in the size of plasmacytomas (by clinical or radiographic examination) for a minimum of 6 weeks, No increase in size or number of lytic bone lesions (development of compression fracture does not exclude response).
Time Frame: Up to 12 cycles of 3 weeks each
Population: mITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 0 | 1

5. Primary Outcome: Number of Participants With Partial Response (PR) as Last Observed Response (LOR)
Description: as for outcome 3
Time Frame: Up to 12 cycles of 3 weeks each
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 0 | 1

6. Primary Outcome: Number of Participants With Stable Disease (SD) as Best Response (BR)
Description: Stable disease included not meeting the criteria for MR or PD.
Time Frame: Up to 12 cycles of 3 weeks each
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 3 | 4

7. Primary Outcome: Number of Participants With Stable Disease (SD) as Last Observed Response (LOR)
Description: Stable disease included not meeting the criteria for MR or PD.
Time Frame: Up to 12 cycles of 3 weeks each
Population: mITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 2 | 4

8. Primary Outcome: Number of Participants With Progressive Disease (PD) PD as Best Response (BR)
Description: PD includes one or more of the following criteria: >25% increase in the level of serum monoclonal paraprotein, which must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation, >25% increase in 24 hr urinary light chain excretion, which must also be an absolute increase of at least 200 mg/24 hr and confirmed on a repeat investigation, >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10%., Definite increase in the size of existing lytic bone lesions or soft tissue plasmacytomas, Development of new bone lesions or soft tissue plasmacytomas (not including compression fracture), Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.8 mmol/L not attributable to any other cause).
Time Frame: Up to 12 cycles of 3 weeks each
Population: mITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 1 | 2

9. Primary Outcome: Number of Participants With Progressive Disease (PD) PD as Last Observed Response (LOR)
Description: as for outcome 8
Time Frame: Up to 12 cycles of 3 weeks each
Population: mITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Participants | 2 | 4

10. Primary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from first dose until objective tumor progression. Participants who did not experience tumor progression were censored at their last known date in the study. It was estimated using Kaplan-Meier methodology. Participants who did not experience tumor progression were censored at their last known date in the study. The first quartile for time to disease progression was evaluated when 25th percentile of participants of mITT population reported disease progression. Similarly, median and 75th percentile of participants of MITT population was planned to be reported. If, less than 75th percentile of participants reported disease progression at the end of the study period, then the observation was censored for the purpose of this analysis and in such case the data was planned to be reported as not evaluable (NA).
Time Frame: From Day 1 till disease progression (approximately 12 cycles of 3 weeks each)
Population: mITT Population. Only those participants available at the specified timepoints were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 4 | 9
Months | 2.8 [2.0 to 2.8] | 2.8 [1.3 to NA] — NA indicates 'Q3 is not evaluable' as less than 75th percentile of participants reported disease progression.

11. Primary Outcome: Change From Baseline in Hematology: White Blood Cell (WBC) Count, Neutrophils, Lymphocytes, Platelets
Description: Blood samples collected to evaluate the hematology parameters were WBC count, neutrophils, lymphocytes and platelets. Change from Baseline was defined as the value of Baseline minus from the End of study visit. Baseline was defined as Day 1.
Time Frame: Baseline (Day 1) and End of Study assessments/follow-up approximately 28 days (+/- 7 days) following the last dose of SRT501 or SRT501 and bortezomib (approximately 280 days)
Population: Safety Population. Only those participants available at the specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (L)
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 24 | 9
10^9 cells per liter (L)
  WBC count: number analyzed (Participants) | 21 | 9
  WBC count | 0.55 (2.76) | 0.07 (1.48)
  Neutrophils: number analyzed (Participants) | 21 | 9
  Neutrophils | 0.27 (1.32) | 0.32 (1.46)
  Lymphocytes: number analyzed (Participants) | 21 | 9
  Lymphocytes | 0.09 (1.30) | -0.34 (0.30)
  Platelets: number analyzed (Participants) | 21 | 9
  Platelets | -12.1 (58.1) | -9.3 (66.3)

12. Primary Outcome: Change From Baseline in Hematology: Hematocrit
Description: Blood samples were collected to evaluate the hematology parameter hematocrit. Change from Baseline was defined as the value of baseline minus from the End of study visit. Baseline was defined as Day 1.
Time Frame: as for outcome 11
Population: Safety population. Only those participants available at the specified time-points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 21 | 9
Proportion of red blood cells in blood | -0.04 (0.05) | -0.03 (0.04)

13. Primary Outcome: Change From Baseline in Hematology: Hemoglobin
Description: Blood samples were collected to evaluate the hematology parameter hemoglobin. Change from Baseline was defined as the value of Baseline minus from the End of study visit. Baseline was defined as Day 1.
Time Frame: as for outcome 11
Population: Safety population. Only those participants available at the specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per litre
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 21 | 9
Gram per litre | -11.4 (15.0) | -9.17 (14.3)

14. Primary Outcome: Change From Baseline in Hematology: Red Blood Cell (RBC)
Description: Blood samples were collected to evaluate the hematology parameter RBC. Change from Baseline was defined as the value of Baseline minus from the End of study visit. Baseline was defined as Day 1.
Time Frame: as for outcome 11
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 21 | 9
10^12 cells per liter | -0.30 (0.51) | -0.16 (0.43)

15. Primary Outcome: Change From in Baseline Biochemistry: Serum Creatinine, Total Bilirubin
Description: Blood samples were collected to evaluate hematology parameters serum creatinine and total bilirubin. Change from Baseline was defined as the value of baseline minus from the End of study visit. Baseline was defined as Day 1.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromole per liter
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 24 | 9
Micromole per liter
  Serum creatinine: number analyzed (Participants) | 20 | 9
  Serum creatinine | 59.8 (123.5) | 3.60 (8.41)
  Total bilirubin: number analyzed (Participants) | 19 | 9
  Total bilirubin | 1.6 (5.65) | 0.80 (2.44)

16. Primary Outcome: Change From Baseline in Biochemistry -Urea, Bicarbonate
Description: Blood samples were collected to evaluate the biochemistry parameter urea and bicarbonate. Change from Baseline was defined as the value of Baseline minus from the End of study visit. Baseline was defined as Day 1.
Time Frame: as for outcome 11
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimole per liter
Groups:
- SRT501 Monotherapy: The eligible participants in this arm received 5 g of SRT501, orally every morning at the same time approximately 15-30 minutes following consumption of breakfast) on all dosing days, for 20 consecutive days in a 21-day cycle for a maximum period of 12 cycles. There was no time between the cycles i.e Day 1 of a cycle was started on the day following Day 21 of the previous cycle. SRT501 was not administered on Day 21 of each cycle.
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 24 | 9
millimole per liter
  Bicarbonate: number analyzed (Participants) | 14 | 7
  Bicarbonate | -0.81 (3.41) | 0.64 (1.10)
  Urea: number analyzed (Participants) | 20 | 9
  Urea | 3.50 (7.87) | -0.18 (1.61)

17. Primary Outcome: Change From Baseline in Biochemistry: Prothrombin Time (PT)/ International Normalized Ratio (INR)
Description: Blood samples were collected to evaluate the biochemistry parameter PT/INR. Change from Baseline was defined as the value of Baseline minus from the End of study visit. Baseline was defined as Day 1.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants available at the particular timepoints were analyzed
Measure: Mean (Standard Deviation); unit: Ratio of PT/INR
Groups:
- SRT501 + Bortezomib: The eligible participants in this arm received an intravenous solution of Bortezomib at 1.3 mg/m^2 in conjunction with SRT501 (5.0 g/day) daily dosing. Bortezomib was administered prior to breakfast and SRT501 administration, on Day 1, 4, 8 and 11 in every 21 day cycle. It was given as per the local institution's guidelines and standards of care.SRT501 + Bortezomib, is a subset of arm SRT501 monotherapy.
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 13 | 6
Ratio of PT/INR | 0.11 (0.41) | 0.05 (0.16)

18. Secondary Outcome: Plasma Concentrations of SRT501 at Indicated Time Points
Description: Pharmacokinetic sampling on Day1/2 and Day 20/21 of Cycle 1 for participants ready to participate was planned. The sampling was planned to be collected at timepoints on Cycle 1 Day 1 at pre-dose, 30 minute, 1 hour, 2 hour, 4 hour, 6 hour and 24 hour post-dose and the same timepoints on Day 2 and Day 20 post- dose. It was to be collected in participants who fasted atleast for an hour. Due to early termination of the study, the data for Pharmacokinetic analysis was not collected.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 2 and Cycle 1 Day 20 at pre-dose, 30 minute, 1 hour, 2 hour, 4 hour, 6 hour and 24 hour post-dose. Day 2 and Day 20, samples collected post-dose. Each cycle duration was 21 days.
Population: Subjects who receive study drug and have adequate pharmacokinetic data available will be included in the pharmacokinetics population, with data summarized by dose group. Data not collected due to early termination of the study.
Groups:
- SRT501 Monotherapy: The eligible participants in this arm received 5 g of SRT501, oral suspension every morning at the same time approximately 15-30 minutes following consumption of breakfast) on all dosing days, for 20 consecutive days in a 21-day cycle for a maximum period of 12 cycles. There was no time between the cycles i.e Day 1 of a cycle was started on the day following Day 21 of the previous cycle. No administration of SRT501, will occur on Day 21 of each cycle.
Arm/Group | SRT501 Monotherapy | SRT501 + Bortezomib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 to Follow up (Approximately up to 12 cycles of 3 weeks each)
Description: SAE and Non-serious data was reported for safety population. At the time the participant was judged to have progressive disease (PD) (after receiving at least 4 cycles of SRT501 monotherapy), the participant also received bortezomib (1.3 mg/m2 on Day 1, Day 4, Day 8, and Day 11 in a 21 day cycle) in conjunction with daily SRT501 dosing (N=9). Data presented for SRT501, which combines AE details for SRT501 as well as SRT501 and Bortezomib.
Groups:
- SRT501: The eligible participants in this arm received 5 g of SRT501, oral suspension every morning at the same time approximately 15-30 minutes following consumption of breakfast) on all dosing days, for 20 consecutive days in a 21-day cycle for a maximum period of 12 cycles. There was no time between the cycles i.e Day 1 of a cycle was started on the day following Day 21 of the previous cycle. No administration of SRT501, will occur on Day 21 of each cycle.
Arm/Group | SRT501
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 12/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRT501 (N=24)
Anemia (Blood and lymphatic system disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Pyrexia (General disorders) | 2
Pneumonia (Infections and infestations) | 2
Neutropenic sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Renal failure acute (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SRT501 (N=24)
Nausea (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 11
PYREXIA (General disorders) | 4
OEDEMA PERIPHERAL (General disorders) | 3
CHILLS (General disorders) | 2
DISEASE PROGRESSION (General disorders) | 2
HEADACHE (Nervous system disorders) | 9
NEUROPATHY PERIPHERAL (Nervous system disorders) | 6
DIZZINESS (Nervous system disorders) | 5
DYSGEUSIA (Nervous system disorders) | 2
LETHARGY (Nervous system disorders) | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 6
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2
ANOREXIA (Metabolism and nutrition disorders) | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
NASOPHARYNGITIS (Infections and infestations) | 2
ORAL CANDIDIASIS (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 2
RHINITIS (Infections and infestations) | 2
URINARY TRACT INFECTION (Infections and infestations) | 2
ANAEMIA (Blood and lymphatic system disorders) | 8
NEUTROPENIA (Blood and lymphatic system disorders) | 6
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2
DEPRESSION (Psychiatric disorders) | 4
CONFUSIONAL STATE (Psychiatric disorders) | 3
ANXIETY (Psychiatric disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 4
WEIGHT DECREASED (Investigations) | 3
BLOOD CREATININE INCREASED (Investigations) | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 2
HYPERTENSION (Vascular disorders) | 3
TACHYCARDIA (Cardiac disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Eructation (Gastrointestinal disorders) | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
The study of Multiple Myeloma, was terminated early due to minimal efficacy signal observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.